CLINICAL TRIAL: NCT00967681
Title: Efficacy and Safety of Nutritional Supplement ONCOXIN in Patients With Breast Fibrocystic Disease
Brief Title: Efficacy and Safety of ONCOXIN in Patients With Breast Fibrocystic Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAT-0901-CU
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Breast Fibrocystic Disease
MeSH Terms: conditions — Fibrocystic Breast Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Oncoxin, a nutritional supplement
  Interventions: Dietary Supplement: Oncoxin
- B (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oncoxin — (caplets 300 mg), three oral caplets per day for 24 weeks
  Arms: A
Dietary Supplement: Placebo — (caplets 300 mg), three oral caplets per day for 24 weeks
  Arms: B

SUMMARY:
The purpose of the study is to evaluate whether Oncoxin, a nutritional supplement, improves the clinical and ultrasonographic results in comparison with placebo during 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and ultrasonographic confirmation of breast fibrocystic disease.
* Patients older than 20 years.
* Female patients.
* Informed consent.

Exclusion Criteria:

* Presents of another disease not well controlled.
* Pregnant women or lactating.
* Patient which are receiving another products from other investigations trials.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The ultrasonographic improvement at 24 weeks (end of the treatment) | 24 weeks
Adverse effects at 24 weeks (end of the treatment) | 24 weeks

SECONDARY OUTCOMES:
Lesion size according clinical measurement at 24 weeks (end of the treatment) | 24 weeks
Pain according patient examination at 24 weeks (end of the treatment) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daisy Hernández, MD, Principal Investigator — Ramón González Coro Hospital
Locations (1):
- "Ramón González Coro" Gynecologic and Obstetric Hospital, Havana, La Habana, Cuba